CLINICAL TRIAL: NCT02693626
Title: The Efficacy of Mobile Phone-based Text Message Interventions ('Happy Quit') for Smoking Cessation in China
Brief Title: Happy Quit for Smoking Cessation in China
Acronym: HQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Purdue University (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Dr., Central South University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2015S007
Record Dates: First submitted 2016-02-19; First posted 2016-02-29 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2018-04

CONDITIONS: Smoking Cessation
Keywords: mobile phone-based text message interventions; 'Happy Quit'; smoking cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- intensive cessation message (Experimental): Participants who allocate to this intervention group will receive regular, personalized text messages providing smoking cessation advice, support, and distraction. A quit day will be negotiated with each participant, and one to five messages will be sent per day for the time leading up to the quit day and the following 12 weeks.
  One to three messages will be sent per week until the end of the 24 week follow up. In order to measure the main two outcomes (self-reported continuous smoking abstinence and point prevalence of abstinence), continuous smoking abstinence, point prevalence of abstinence, how many cigarettes per day during the last 4 weeks and past 1 week if they are still smoking, they will also be checked by phone call at 4, 8, 12, 16, 20, 24 week points.
  Interventions: Behavioral: intensive cessation message
- No cessation message intervention (No Intervention): Control group participants only will receive one text message every week, thanking them for being in the study, providing study center contact details, and reminding them of the time until their free month at the end of follow up. Another one to two messages will be sent per week until the end of the 24 week. In order to measure the main two outcomes (self-reported continuous smoking abstinence and point prevalence of abstinence), continuous smoking abstinence, point prevalence of abstinence, how many cigarettes per day during the last 4 weeks and past 1 week if they are still smoking, they will also be checked by phone call at 4, 8, 12, 16, 20, 24 week points.
- Not intensive cessation message (Experimental): Participants who allocate to this intervention group will receive regular, personalized text messages providing smoking cessation advice, support, and distraction. A quit day will be negotiated with each participant, and one to five messages will be sent per week for the time leading up to the quit day and the following 12 weeks.
  One to three messages will be sent per week until the end of the 24 week follow up. In order to measure the main two outcomes (self-reported continuous smoking abstinence and point prevalence of abstinence), continuous smoking abstinence, point prevalence of abstinence, how many cigarettes per day during the last 4 weeks and past 1 week if they are still smoking, they will also be checked by phone call at 4, 8, 12, 16, 20, 24 week points.
  Interventions: Behavioral: Not intensive cessation message

INTERVENTIONS:
Behavioral: intensive cessation message — Mobile phone-based text message （three to five messages per day） interventions ('Happy Quit') for smoking cessation for 12 weeks with 24 week follow up.
  Arms: intensive cessation message
Behavioral: Not intensive cessation message — Mobile phone-based text message （three to five messages per week） interventions ('Happy Quit') for smoking cessation for 12 weeks with 24 week follow up.
  Arms: Not intensive cessation message

SUMMARY:
The primary objective of this proposed three-year (January 01, 2016 to December 31, 2018) project is to assess whether a program of widely accessed mobile phone-based text message interventions ('Happy Quit') will be effective at helping people in China who smoke, to quit. Based on the efficacy of previous studies in smoking cessation, it is hypothesized that 'Happy Quit' will be an effective, feasible and affordable smoking cessation program in China.

DETAILED DESCRIPTION:
Background: Considering the extreme shortage of smoking cessation services in China, and the acceptability, feasibility and efficacy of mobile phone-based text message interventions for quitting smoking in other countries, here a study of "the efficacy of mobile phone-based text message interventions ('Happy Quit') for smoking cessation in China"has been proposed.

Objectives: The primary objective of this proposed three-year (January 01, 2016 to December 31, 2018) project is to assess whether a program of widely accessed mobile phone-based text message interventions ('Happy Quit') will be effective at helping people in China who smoke, to quit. Based on the efficacy of previous studies in smoking cessation, it is hypothesized that'Happy Quit' will be an effective, feasible and affordable smoking cessation program in China.

Methods: In this single-blind, randomized trial, undertaken in China, about 2,000 smokers willing to make a quit attempt will be randomly allocated, using an independent telephone randomization system that includes a minimization algorithm balancing for sex (male, female), age (19-34 or >34 years), educational level (≤ or >12 years), and Fagerstrom score for nicotine addiction (≤5, >5), to 'Happy Quit', comprising motivational messages and behavioral-change support, or to a control group that receives text messages unrelated to quitting.

Outcome measures: The primary outcome will be continuous smoking abstinence. A secondary outcome will be point prevalence of abstinence. Abstinence will be assessed by means of brief telephone interviews at six time points (4, 8, 12, 16, 20 and 24 weeks post-intervention). A third outcome will be reductions in number of cigarettes smoked per day.

Implications: The results will provide valuable insights into bridging the gap between need and services received for smoking cessation interventions and tobacco use prevention in China. It will also serve as mHealth model for extending the public health significance of other interventions, such as mental health interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Daily Chinese cigarette smokers.
2. 18 years of age and older living.
3. Being able to read and write in Chinese.
4. Owning a text-capable cell phone and knowing how to text.
5. Willing to make an attempt to quit smoking in the next month.
6. Willing to provide informed consent to participate in the study.

Exclusion Criteria:

1. Nonsmokers
2. Below 18 years old.
3. Unable to read and write in Chinese.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1369 (Actual)
Dates: Start 2016-08-17 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be self-reported and biologically verified continuous smoking abstinence. | Six month

SECONDARY OUTCOMES:
A secondary outcome will be point prevalence of abstinence. | six month

IPD SHARING:
Plan to Share IPD: Yes
I would be happy to share the data with everyone.

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Liao Y, Wu Q, Kelly BC, Zhang F, Tang YY, Wang Q, Ren H, Hao Y, Yang M, Cohen J, Tang J. Effectiveness of a text-messaging-based smoking cessation intervention ("Happy Quit") for smoking cessation in China: A randomized controlled trial. PLoS Med. 2018 Dec 18;15(12):e1002713. doi: 10.1371/journal.pmed.1002713. eCollection 2018 Dec. PMID 30562352
- [Derived] Liao Y, Wu Q, Tang J, Zhang F, Wang X, Qi C, He H, Long J, Kelly BC, Cohen J. The efficacy of mobile phone-based text message interventions ('Happy Quit') for smoking cessation in China. BMC Public Health. 2016 Aug 19;16(1):833. doi: 10.1186/s12889-016-3528-5. PMID 27543164
- Available data/document: Study Protocol: 15OCCSULiaoYanhui — http://pan.baidu.com/disk/home#list/path=%2F — Please send me email: tangliaoyanhui@163.com if you cannot open it.